CLINICAL TRIAL: NCT07002073
Title: Comparison of the Hemodynamic Effects of Ketamine - Dexmedetomidine (Ketodex) Versus Propofol-ketamine Admixture (Ketofol) During Induction of Anesthesia in Elderly: A Randomized Comparative Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Emad Mohamed Ahmed Abdelhafez, Lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-451-2024
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Ketamine-dexmedetomidine Induction of Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine-dexmedetomidine admixture induction of Anesthesia (Active Comparator): Intravenous Induction of Anesthesia Using a Mixture of Ketamine and dexmedetomidine in a ratio of 1 mg ketamine to 0.5 ug dexmedetomidine given in a dose of 1mg/kg ketamine and 0.5 ug/kg dexmedetomidine to elderly patients
  Interventions: Drug: Intravenous Induction of Anesthesia
- propofol - ketamine admixture induction of Anesthesia (Active Comparator): Intravenous Induction of Anesthesia Using a Mixture of Ketamine and Propofol in a ratio of 1:1 in elderly patients given in a dose of 1 mg/kg ketamine and 1 mg/kg propofol
  Interventions: Drug: Intravenous Induction of Anesthesia

INTERVENTIONS:
Drug: Intravenous Induction of Anesthesia — To compare incidence of hypotension following ketodex versus ketofol during intavenous induction of general anesthesia in elderly patients
  Other Names: Effect of drug mixtures on hypotension during induction of Anesthesia in elderly patients

SUMMARY:
To compare the hemodynamic effects of Ketamine-Dexmedetomidine admixture (Ketodex) versus propofol-ketamine admixture (Ketofol) during induction of anesthesia in elderly

DETAILED DESCRIPTION:
This study details the protocol for anesthetic induction and maintenance, allocating patients into Ketodex (KD) and Ketofol (KP) groups. Prior to anesthesia, a fluid challenge (4 mL/kg over 10 minutes) was administered to assess volume status, with repeated challenges until pulse pressure increased by less than 15% of baseline. For induction, all patients received 1 mg/kg lidocaine. KD patients then received 1 mg/kg ketamine + 0.5 µg/kg dexmedetomidine over 10 minutes, while KP patients received 0.15-0.20 mL/kg of a ketofol admixture. Loss of consciousness, defined by no response to auditory commands and absent eyelash reflex, led to the administration of 0.6 mg/kg rocuronium. After 2 minutes of mask ventilation, an endotracheal tube was inserted. Anesthesia was maintained with isoflurane (0.9-1% end-tidal), and Ringer's lactate solution was infused at 4 mL/kg/hour. Hemodynamic stability was rigorously managed: hypotension (mean blood pressure (MBP) ≤ 80% of baseline and/or MBP < 60 mmHg) occurring up to 15 minutes post-intubation or skin incision was treated with 5 µg norepinephrine boluses, repeatable every 2 minutes. Severe post-induction hypotension (MBP ≤ 60% of baseline) prompted 5 µg norepinephrine boluses every minute, with 1-minute interval blood pressure monitoring. Hypertension (mean arterial pressure > 120% of baseline) was managed with 0.25 mg/kg IV propofol, while bradycardia (heart rate < 45 bpm) was treated with 0.5 mg IV atropine. Blood pressure and heart rate were continuously monitored at specified intervals, with subsequent hemodynamic management left to the discretion of the attending anesthetist after 15 minutes post-intubation or skin incision.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (>65 years)
* ASA physical status I-III
* Elective non-cardiac surgery under general anesthesia.

Exclusion Criteria:

* Patients with severe cardiac morbidities (impaired contractility with ejection fraction < 50%, heart block, arrhythmias, tight valvular lesions, metabolic equivalent [MET] less than 4
* Patients on angiotensin-converting enzyme inhibitors and angiotensin receptor blockers medications
* Patients with uncontrolled hypertension
* patients undergoing adrenalectomy
* patients with body mass index <18 or > 35 kg/m²
* patient with allergy to any of the study drugs.
* patient is considered to be a difficult intubation in the preoperative assessment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-induction hypotension | 12 months
  Incidence of post-induction hypotension (MBP ≤80% of baseline or <60 mmHg) during the period from induction of anesthesia until 16-minutes after intubation providing that skin incision will be after 16-minutes interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals, Cairo, Giza Governorate, Egypt